CLINICAL TRIAL: NCT05358665
Title: An Investigation of Temporomandibular Pain, Headache, and Fatigue in Relation With Long-Term Mask Use During the Pandemics
Brief Title: The Effects of Long-Term Mask Use in the Pandemic Period
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-586/58
Record Dates: First submitted 2022-04-28; First posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: COVID-19
Keywords: mask; temporomandibular joint disorders; headache; fatigue
MeSH Terms: conditions — COVID-19; Temporomandibular Joint Disorders; Headache; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: There are individuals who use masks for less than 4 hours daily.
  Interventions: Other: mask use
- Group 2: There are individuals who use masks for 4-8 hours daily.
  Interventions: Other: mask use
- Group 3: There are individuals who use masks for more than 8 hours daily.
  Interventions: Other: mask use

INTERVENTIONS:
Other: mask use — long term mask use

SUMMARY:
Various restrictions have been made all over the world due to coronavirus pandemics. In addition to situations such as social isolation and hygiene, the use of masks is among these rules. In addition to the protection it provides, the use of masks causes some negative situations in individuals. For this reason, the aim of our study is to examine the effects of long-term mask use on temporomandibular dysfunction, headache and fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* Able to read and understand
* Volunteer to participate

Exclusion Criteria:

* Malignity history
* Head/Face surgery history

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People using masks
Sampling Method: Non-Probability Sample
Enrollment: 909 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Temporomandibular Dysfunction | Baseline
  According to the scores obtained from the scale, 0-15 points mean no temporomandibular dysfunction symptoms, 20-45 points mean mild temporomandibular dysfunction symptoms, 50-65 points mean moderate temporomandibular dysfunction symptoms, and 70-100 severe temporomandibular dysfunction symptoms.

SECONDARY OUTCOMES:
Mask Use Symptoms | Baseline
  It was evaluated whether long-term use of masks had negative effects such as pain, skin problems, sleep, voice problems, temporomandibular problems. The results are given in terms of frequency.
Perceptions of Mask Use | Baseline
  The mask discomfort perception scale was used to evaluate the uncomfortable perceptions of mask use over visual analog scale. Scores were recorded as 0- no problem, 10- many problems.
Fatigue | Baseline
  Fatigue was assessed with the Chalder Fatigue Scale. Each item in the scale consisting of physical and mental fatigue sub-parameters is scored between 0-3. The total score ranges from 0 to 33, and as the score increases, fatigue increases.
Type of Headache | Baseline
  Individuals were asked to show the localization of the headache they experienced through the presented figures.
Trigger point of temporomandibular joint | Baseline
  Pain intensity at the temporomandibular joint trigger points was evaluated with visual analog scale. It was recorded as 0, no pain; 10 very severe pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yildirim Beyazit University, Ankara, Turkey (Türkiye)